CLINICAL TRIAL: NCT03351426
Title: Neuromodulation With Transcranial Direct Current Stimulation (tDCS) to Control Excess Weight
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Pedro de la Villa Polo, Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEI/HU/2016/11
Record Dates: First submitted 2017-11-15; First posted 2017-11-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Overweight and Obesity
Keywords: obesity; overweight; neuromodulation; transcranial direct current stimulation (tDCS)
MeSH Terms: conditions — Overweight; Obesity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The study is double blind. Neither the participants or the investigator delivering the intervention and collecting the outcomes will be aware of the group allocation. This is achieved via sham tDCS procedure and blinding of tDCS parameters with code system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS Group (Active Comparator): Subjects will receive a total of eight tDCS sessions: 1st week five daily sessions (Monday to Friday), followed by 2nd week three sessions only (Monday, Wednesday, Friday). tDCS sessions will consist of 20 minutes stimulation at 2mA. Target: left dorsolateral prefrontal cortex (DLPFC). Montage: 5x5 sponge electrodes placed over EEG 10:20 system location F3 (anode) and right supraorbital area (cathode).
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS Group (Sham Comparator): Subjects will receive a total of eight tDCS sessions: 1st week five daily sessions (Monday to Friday), followed by 2nd week three sessions only (Monday, Wednesday, Friday). tDCS sessions will be sham stimulation (30-second ramp up and down). Target: left dorsolateral prefrontal cortex (DLPFC). Montage: 5x5 sponge electrodes placed over EEG 10:20 system location F3 (anode) and right supraorbital area (cathode).
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — Transcranial Direct Current Stimulation (tDCS) is a noninvasive form of neuromodulation that uses constant, low-intensity direct current delivered via electrodes that are placed on the head.

SUMMARY:
The purpose of this study is to examine the effects of noninvasive neuromodulation with transcranial direct current stimulation (tDCS) aimed at enhancing the excitability of the left prefrontal cortex in middle-aged women with excess body weight. This is a randomized, parallel, double-blind study with a duration of 4 weeks. Outcome measures will include changes in performance in a computerized task assessing executive functions, subjective measures of food craving and appetite and changes in body weight.

DETAILED DESCRIPTION:
A total of 40 subjects with overweight or class I obesity will be enrolled and randomized into either Group 1) Active tDCS or Group 2) Sham (control) tDCS. The duration of the study will be 4 weeks. During the first two weeks participants will receive eight sessions of tDCS. At week 2 they will also start a hypocaloric diet. The stimulation sessions (duration: 20 minutes, intensity: 2 mA) will be applied once daily (5 days in a row) during the first week and 3 alternate days (Monday, Wednesday and Friday) during the second week. At week 2 and until the end of the study subjects will also start a hypocaloric diet.

The study aims are:

1. To examine whether anodal tDCS applied over the left prefrontal cortex can improve executive functions/inhibitory control and reduce subjective ratings of food craving and appetite.
2. To study whether anodal tDCS applied over the left prefrontal cortex, in combination with a hypocaloric diet, can facilitate weight reduction and maintenance over time.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 25 and 35 kg/m2

Exclusion Criteria:

* Endocrinology disorder, such as diabetes mellitus or thyroid disease
* Addiction
* Neurological, psychiatric or any other major medical condition
* Hormonal therapy
* Contraindications to receive tDCS (past history of seizures or epilepsy, metallic implants on the head, skin disease or lesions in the area to be stimulated).

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Body weight | Baseline, 4 weeks (end of the study)
  Change

SECONDARY OUTCOMES:
Appetite (hunger) | Baseline, 4 weeks (end of the study)
  Change, evaluated via visual analogue scale (VAS). Self-reported scores to the question "How hungry are you?" representing the current state of the participant will be assessed with a horizontal line, 100 mm in length, anchored by the word descriptors "Not at all" and "Extremely", following standard methods, based on Blundell et al 2009.
Food craving | Baseline, 4 weeks (end of the study)
  Change, evaluated via scores in the State Food Craving Questionnaire developed by Cepeda-Benito (Moreno et al 2008).

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Médico Complutense, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Val-Laillet D, Aarts E, Weber B, Ferrari M, Quaresima V, Stoeckel LE, Alonso-Alonso M, Audette M, Malbert CH, Stice E. Neuroimaging and neuromodulation approaches to study eating behavior and prevent and treat eating disorders and obesity. Neuroimage Clin. 2015 Mar 24;8:1-31. doi: 10.1016/j.nicl.2015.03.016. eCollection 2015. PMID 26110109
- [Background] Gluck ME, Alonso-Alonso M, Piaggi P, Weise CM, Jumpertz-von Schwartzenberg R, Reinhardt M, Wassermann EM, Venti CA, Votruba SB, Krakoff J. Neuromodulation targeted to the prefrontal cortex induces changes in energy intake and weight loss in obesity. Obesity (Silver Spring). 2015 Nov;23(11):2149-56. doi: 10.1002/oby.21313. PMID 26530931
- [Background] Truong DQ, Magerowski G, Blackburn GL, Bikson M, Alonso-Alonso M. Computational modeling of transcranial direct current stimulation (tDCS) in obesity: Impact of head fat and dose guidelines. Neuroimage Clin. 2013 May 31;2:759-66. doi: 10.1016/j.nicl.2013.05.011. eCollection 2013. PMID 24159560
- [Background] Alonso-Alonso M. Translating tDCS into the field of obesity: mechanism-driven approaches. Front Hum Neurosci. 2013 Aug 27;7:512. doi: 10.3389/fnhum.2013.00512. eCollection 2013. PMID 23986687
- [Background] Heinitz S, Reinhardt M, Piaggi P, Weise CM, Diaz E, Stinson EJ, Venti C, Votruba SB, Wassermann EM, Alonso-Alonso M, Krakoff J, Gluck ME. Neuromodulation directed at the prefrontal cortex of subjects with obesity reduces snack food intake and hunger in a randomized trial. Am J Clin Nutr. 2017 Dec;106(6):1347-1357. doi: 10.3945/ajcn.117.158089. Epub 2017 Oct 18. PMID 29046305
- [Background] Ljubisavljevic M, Maxood K, Bjekic J, Oommen J, Nagelkerke N. Long-Term Effects of Repeated Prefrontal Cortex Transcranial Direct Current Stimulation (tDCS) on Food Craving in Normal and Overweight Young Adults. Brain Stimul. 2016 Nov-Dec;9(6):826-833. doi: 10.1016/j.brs.2016.07.002. Epub 2016 Jul 15. PMID 27498606
- [Background] Macedo IC, de Oliveira C, Vercelino R, Souza A, Laste G, Medeiros LF, Scarabelot VL, Nunes EA, Kuo J, Fregni F, Caumo W, Torres ILS. Repeated transcranial direct current stimulation reduces food craving in Wistar rats. Appetite. 2016 Aug 1;103:29-37. doi: 10.1016/j.appet.2016.03.014. Epub 2016 Mar 10. PMID 26972354
- [Background] Stoeckel LE, Birch LL, Heatherton T, Mann T, Hunter C, Czajkowski S, Onken L, Berger PK, Savage CR. Psychological and neural contributions to appetite self-regulation. Obesity (Silver Spring). 2017 Mar;25 Suppl 1(Suppl 1):S17-S25. doi: 10.1002/oby.21789. PMID 28229541
- [Background] Moreno S, Rodriguez S, Fernandez MC, Tamez J, Cepeda-Benito A. Clinical validation of the trait and state versions of the Food Craving Questionnaire. Assessment. 2008 Sep;15(3):375-87. doi: 10.1177/1073191107312651. Epub 2008 Feb 29. PMID 18310596
- [Background] Blundell J, deGraaf K, Finlayson G, Halford JCG, Hetherington M, King N, et al., Chapter 8. Measuring food intake, hunger, satiety, and satiation in the laboratory, in: Allison DB and Baskin ML, (Eds.), Handbook of assessment methods for eating behaviors and weight-related problems: measures, theory, and researched, SAGE Publications, Inc, Thousand Oaks, CA, 2009.